CLINICAL TRIAL: NCT05484570
Title: Natural History Study for DNA Repair Disorders
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUR-2022-30942
Record Dates: First submitted 2022-07-12; First posted 2022-08-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: DNA Repair Disorder; Cockayne Syndrome; Xeroderma Pigmentosum; Trichothiodystrophy
MeSH Terms: conditions — DNA Repair-Deficiency Disorders; Cockayne Syndrome; Xeroderma Pigmentosum; Trichothiodystrophy Syndromes | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Comprehensive metabolic panel (CMP) that includes electrolytes, ALT, AST, and LDH.
  2. GGT
  3. Bilirubin
  4. Complete blood count (CBC)
  5. Neurofilament light (NfL)40-42
  6. Glial fibrillary acidic protein (GFAP)43
  7. Total tau (t-tau)44
  8. Ubiquitin C-terminal hydrolase (UCHL1)45
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosed: Patients who are diagnosed with a DNA Repair Disorder
  Interventions: Other: Interval History; Other: Physical Examination; Other: ECAB Assessment; Other: Gait Assessment; Other: Specimen Sample Collection
- Control: Healthy family members of enrolled diagnosed participants.
  Interventions: Other: ECAB Assessment; Other: Gait Assessment; Other: Specimen Sample Collection

INTERVENTIONS:
Other: Interval History — The study coordinator or another team member will review standard health questions relevant to DNA repair disorders. The control group will not undergo an interval history. These questions will include:
  1. How the participant's appetite and general weight trajectory has been since the last assessment
  2. Any episodes of unexplained bleeding or bruising
  3. Any jaundice
  4. General level of alertness and interaction with family and others
  5. Any changes in cognitive function such as speech, following commands, comprehension
  6. Any changes in motor function, including the development of tremors and stiffness in movements
  Groups: Diagnosed
Other: Physical Examination — A board-certified neurologist (the principal investigator) will perform a general physical examination and a neurological examination and complete a standard CRF to document relevant findings. The control group will not undergo a physical examination.
  Groups: Diagnosed
Other: ECAB Assessment — An Early Clinical Assessment of Balance (ECAB) will be performed by the physical therapist. Part I can be assessed in all affected individuals, and Part II requires ambulation. For non-ambulatory individuals, only Part I will be applied. The items in the ECAB are summarized as follows:
  Part I. Head and trunk postural control (maximum 36 points) Head righting - lateral (right and left) Head righting - extension Head righting - flexion Rotation in trunk (right and left) Equilibrium reactions in sitting (right and left) Protective extension - side Protection extension - backward Part II. Sitting and standing postural control (maximum 64 points) Sitting with back unsupported but feet supported on floor or on a stool Sitting to standing Standing unsupported with eyes closed Standing unsupported with feet together Turns 360 degrees Placing alternate foot on the step while standing unsupported
Other: Gait Assessment — For ambulatory participants, the physical therapist will also assess standardized gait outcome measures, including:
  1. Gait Speed: may be measured over a 10 meter distance, assessing both "comfortable" walking speed and "fast" walking speed
  2. 10-meter walk/run: timed assessment at fastest gait attainable. This assessment would be omitted for those participants who are determined to have a high fall risk.
  3. Timed Up and Go (TUG): time to stand from a chair, walk 3 meters, go around a cone, and return to the chair (with or without an assistive device)
  4. Dynamic Gait Index (DGI): assesses 8 balance challenges while walking
Other: Specimen Sample Collection — Total blood volumes collected at each visit will be limited to 5mL/kg body weight, with a maximum of 18mL.
  Saliva samples may be obtained if research is taking place where blood samples cannot be drawn or transferred.

SUMMARY:
This will be a single-center, single-arm, non-interventional natural history study to evaluate the longitudinal clinical course, functional outcome measures, and candidate biomarkers for individuals with DNA repair disorders, including Cockayne syndrome (CS), xeroderma pigmentosum (XP), and trichothiodystrophy (TTD).

DETAILED DESCRIPTION:
This will be a single-center, single-arm, non-interventional natural history study to evaluate the longitudinal clinical course, functional outcome measures, and candidate biomarkers for individuals with DNA repair disorders, including Cockayne syndrome (CS), xeroderma pigmentosum (XP), and trichothiodystrophy (TTD). Our hypothesis is that a reliable and reproducible baseline natural history course can be established for DNA repair disorders using the Early Childhood Assessment of Balance (ECAB) as a primary endpoint and other measures as secondary and exploratory endpoints that may be used in future therapeutic clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cockayne syndrome (CS), xeroderma pigmentosum (XP), or trichothiodystrophy (TTD), based on genetic testing and/or key clinical characteristics l characteristics
* Has one or more of the following neurodevelopmental or neurological complications
* Gross motor delay (non-ambulatory or started walking after age 18 months)
* Language delay (non-verbal or started talking after 18 months)
* Altered muscle tone (hypertonia, dystonia, hypotonia)
* Gait difficulties, including stiff gait, short stride, frequent falls, use of orthotics, use of walker
* Tremors
* Microcephaly
* Is a family member of an individual with the above condition
* No restrictions regarding current ambulatory status
* Minimum age for enrollment eligibility will be 6 months due to fragility of neonates with severe forms of DNA repair disorders and limitations of motor assessment scales in infants younger than 6 months. There will be no maximum age for enrollment eligibility.
* No restrictions regarding gender, race, or ethnicity.
* Voluntary written consent from the participant if adult capable of consenting or parent/guardian if minor or not capable of consenting
* Written consent of Legally Authorized Representative if enrolling adult lacks capacity to consent

Exclusion Criteria:

* Any prior history of systemic gene or cell-based therapy
* Current participation in an interventional clinical trial

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any person 6 months or older who is either diagnosed with a DNA repair disorder, or has a family member who is diagnosed with a DNA repair disorder
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal stability of cerebellar and gait function on neurological examination | 3 years
  The longitudinal stability of cerebellar and gait function will be assessed by the presence or absence of tremors (absence = 1, presence = 0), dysmetria (absence = 1, presence = 0), dysdiadochokinesia (absence = 1, presence = 0) and Gowers sign (absence = 1, presence = 0). The scores will be added to yield a total score ranging from 0 to 4, with 4 representing the best performance.
Longitudinal stability of motor function using gait speed measurement | 3 years
  Longitudinal stability of motor function in study participants as assessed by gait speed measured over a 10 meter distance
Longitudinal stability of motor function using 10 meter walk/run test | 3 years
Longitudinal stability of motor function using Timed Up and Go (TUG) test | 3 years
Longitudinal stability of motor function using the Dynamic Gait Index (DGI) | 3 years

OTHER OUTCOMES:
Exploratory | 3 years
  We have selected the following 4 biomarkers to be measured in serum samples at each study visit:
  1. Neurofilament light (NfL)
  2. Glial fibrillary acidic protein (GFAP)
  3. Total tau (t-tau)
  4. Ubiquitin C-terminal hydrolase (UCHL1)
  We have selected the following 4 biomarkers to be measured in serum samples at each study visit:
  1. Neurofilament light (NfL)40-42
  2. Glial fibrillary acidic protein (GFAP)43
  3. Total tau (t-tau)44
  4. Ubiquitin C-terminal hydrolase (UCHL1)45 To determine whether a serum biomarker can track disease status and progression and serve as a secondary outcome measure. To determine genetic diagnoses for those who are genetically undiagnosed, and to use transcriptomic analyses to seek additional biomarker candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kang, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota- Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will be conducted in accordance with the following publication and data sharing policies and regulations: National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.